CLINICAL TRIAL: NCT01920880
Title: Nociceptive Processing in Acute Cutaneous Nerve Entrapment Syndrome: a Quantitative Sensory Testing Analysis.
Brief Title: Nociceptive Processing in Acute Cutaneous Nerve Entrapment Syndrome
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL43583.091.13
Record Dates: First submitted 2013-07-12; First posted 2013-08-12 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Anterior Cutaneous Nerve Entrapment Syndrome (ACNES)
Keywords: Anterior cutaneous nerve entrapment syndrome; ACNES; chronic abdominal wall pain; CAWP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACNES patients: Patients being treated in past for anterior cutaneous nerve entrapment syndrome
  Interventions: Other: Quantitative Sensory Testing analysis
- Healthy controls: Healthy controls
  Interventions: Other: Quantitative Sensory Testing analysis

INTERVENTIONS:
Other: Quantitative Sensory Testing analysis

SUMMARY:
Rationale: Chronic abdominal pain is a frequently occurring condition. Although hardly ever considered, the abdominal wall is the primary cause in 10-30% of cases. Most often it is caused by entrapment of an intercostal nerve in the anterior rectus sheath, the Anterior Cutaneous Nerve Entrapment Syndrome (ACNES). Treatment consists of local anaesthetic injections combined with methyl-prednisolon. When ineffective, a neurectomy at the site of penetration out of the ventral rectus sheet should be considered. This neurectomy however is effective in 73% of cases, leaving some 25% of patients in pain. Whether these refractory ACNES patients suffer from underlying pathologic pain disorders is subject to investigation, by using quantitative sensory testing (QST).

Objective: To investigate nociceptive processing and possible underlying pathological pain processing mechanisms in ACNES patients.

Study design: An observational case-control study.

Study population: Patients treated for ACNES (n = 50) compared to healthy controls from an existing database.

Measurements: Quantitative sensory testing (QST) of nociception, performed after treatment of ACNES for both successfully treated and refractory patients in comparison to healthy controls. Visual Analogue Scores (VAS) measured before, during and after testing procedures. Pain Anxiety Symptom Scale (PASS) and Pain Catastrophizing Scale (PCS) questionnaires.

Main study parameters: Pressure pain and electrical pain thresholds as investigated by QST. Secondary study parameters are VAS-scores and results of PASS and PCS questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been diagnosed with abdominal complaints, matching ACNES:

   * Patient had a constant site of tenderness that is superficially located with a small (<2cm2) area of maximal tenderness.
   * The most intense pain could be localized with the tip of one finger.
   * Tenderness increased by abdominal muscle tensing (Carnett's test).
2. has been treated (successfully and unsuccessfully) for ACNES.
3. Patient is at least 18 years old on the day the informed consent form will be signed.
4. Patient is willing and able to comply with the trial protocol.
5. Patient is able to speak, read and understand the local language of the investigational site, is familiar with the procedures of the study, and agrees to participate in the study program by giving oral and written informed consent prior to screening evaluations.

Exclusion Criteria:

1. Abdominal complaints were due to a condition other than ACNES (e.g. pain related to scar tissue).
2. Patient has (a history of) another (chronic) pain syndrome that interferes with the interpretation of QST results.
3. Patient has (a history of) Raynaud syndrome or fenomenon, or a medical disorder that interferes with the study measurements or may pose a risk for the patient.
4. Patient does not feel a pinprick test to the lower extremities, due to affected sensory input (e.g. neuropathy as a result of diabetes mellitus).
5. Female patient is pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of ACNES patients that have been treated both successfully and refractory. The control group will consist of demographically equal healthy controls from an existing database
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | > 6 weeks after treatment
  The pressure pain threshold (pPT) will be determined by pressing an electronic pressure algometer, which has a surface area of 1 cm2, on a distinct muscles. The patient will be asked to say 'now' when the sensation is rated as unpleasant. The pressure will be increased at a rate of 50 kPa/sec until the pPT is reached.

SECONDARY OUTCOMES:
Electrical Sensation Threshold (eST) | > 6 weeks after treatment
  Electrical QST will be measured using a computerized electric stimulation device delivering constant current skin stimulation via self-adhesive electrodes.
  Electric sensation threshold (eST): when electric sensation is first felt.
Electrical Pain Threshold (ePT) | > 6 weeks after treatment
  Electrical QST will be measured using a computerized electric stimulation device delivering constant current skin stimulation via self-adhesive electrodes.
  Electric pain threshold (ePT): when electric sensation is rated as unpleasant
Electrical Pain Tolerance Threshold (ePTT) | >6 weeks after treatment
  Electrical QST will be measured using a computerized electric stimulation device delivering constant current skin stimulation via self-adhesive electrodes.
  Electric pain tolerance threshold (ePTT): when electric sensation is intolerable.
Electric Wind-Up Response (e-WUR) | > 6 weeks after treatment
  Electrical QST will be measured using a computerized electric stimulation device delivering constant current skin stimulation via self-adhesive electrodes.
  Electric wind-up response (eWUR): rated pain after repeated stimuli
Visual Analogue Scale | > 6 weeks after treatment
  Patients will be asked to mark on a 100mm VAS line the average pain in a pain diary. The boundaries of these lines are "no pain" on the upper left site and "unbearable pain" on the upper right site.

OTHER OUTCOMES:
Pain and Anxiety Symptom Scale (PASS) | > 6wks after treatment
  The pain anxiety symptom scale measures four aspects of pain related anxiety: 1) fear for pain, 2) cognitive anxiety, 3) flight or avoidance behavior, 4) physiological symptoms of pain. Elevated scores on this 40-item questionnaire indicate a high level of pain- related anxiety.
Pain Catastrophizing Scale (PCS) | > 6wks after treatment
  Pain catastrophizing affects how individuals experience pain. The PCS yields a three component solution comprising ruminating ("I can ́t stop thinking about how much it hurts"), magnifying (e.g. "I'm afraid that something serious might happen"), and helplessness ("There is nothing I can do to reduce the intensity of my pain").
Hospital Anxiety and Depression Scale (HADS) | > 6wks after treatment
  The Hospital Anxiety and Depression Scale is a 14-item questionnaire of which 7 of the items relate to anxiety (HADS-A) and 7 to depression (HADS-D). The scoring system used is a Likert scale (0 to 3 points) and therefore the data returned is ordinal. A patient can score between 0 and 21. The HADS aims to detect emotional disorder in patients under investigation and treatment in medical and surgical departments

CONTACTS AND LOCATIONS:
Overall Officials: H. van Goor, Prof. MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van Rijckevorsel DC, Boelens OB, Roumen RM, Wilder-Smith OH, van Goor H. Treatment response and central pain processing in Anterior Cutaneous Nerve Entrapment Syndrome: An explorative study. Scand J Pain. 2017 Jan;14:53-59. doi: 10.1016/j.sjpain.2016.09.014. Epub 2016 Nov 4. PMID 28850430